CLINICAL TRIAL: NCT05368688
Title: The Role of the Microbiome in Colorectal Cancer Onset and Progression
Brief Title: Microbiome in Colorectal Cancer Onset and Progression
Status: Terminated | Type: Observational
Why Stopped: Recruitment rate was too low to continue the study.
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: V242
Record Dates: First submitted 2022-04-26; First posted 2022-05-10 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer; Tumor; CRC; GI Cancer; Gastrointestinal Cancer
Keywords: Fusobacterium nucleatum; Microbiome; Viome; Biopsy; Intestinal Permeability; Colonoscopy; Surgical resection; stool; urine; saliva; blood
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cancer-free: Have confirmed colorectal cancer-free and Polyp-free colon using colonoscopy
- Pre-cancerous: Have benign or precancerous polyps, including tubulovillous or villous adenomas, using colonoscopy
- Colorectal cancer stage I: Have confirmed TNM staging of colorectal cancer
  The T refers to the size and extent of the main tumor. The main tumor is usually called the primary tumor.
  The N refers to the number of nearby lymph nodes that have cancer. The M refers to whether the cancer has metastasized. This means that the cancer has spread from the primary tumor to other parts of the body.
- Colorectal cancer stage II: Have confirmed TNM staging of colorectal cancer
  The T refers to the size and extent of the main tumor. The main tumor is usually called the primary tumor.
  The N refers to the number of nearby lymph nodes that have cancer. The M refers to whether the cancer has metastasized. This means that the cancer has spread from the primary tumor to other parts of the body.
- Colorectal cancer stage III: Have confirmed TNM staging of colorectal cancer

SUMMARY:
This is an observational study with the goal to improve the robustness of the scientific evidence linking Fusobacterium nucleatum (Fn) and/or other microorganisms to colorectal cancer (CRC) onset and/or progression. This is an approximately three-year study. There are two phases to this study, including: 1) pilot phase, 2) full study. There are also five arms in this study including cancer-free, pre-cancerous, and Colorectal cancer stages (I-III). The pilot study will include the recruitment of 50 participants per group (i.e., total of 250 participants). The full study will have an additional 150 participants per group (total of 1,000 participants). This study will recruit using clinical sites in the United States.

There are 5 timepoints in this study. If the participants are found to be medically eligible through diagnosis and medical information, they will provide samples (including: saliva, blood, urine, stool and tumor biopsy) at each timepoint and during the study. They will also answer health and wellness questions during this study. Additional data collection, including medical data, biopsies and other biological samples might happen at interim timepoints in case of adenoma/cancer disease progression (recurrence, metastasis). The participant's healthcare provider will determine if additional biopsies are required as a part of the standard of care. If collected, additional samples will be sent for research purposes.

DETAILED DESCRIPTION:
This is an exploratory, longitudinal study that will follow approximately 1,000 participants over 4-6 clinical sites nationwide over a period of 3-4 years and collect molecular and phenotype data to obtain insights into the microbiome and colorectal cancer. Each site will enroll approximately 166-250 participants in total. Those that are polyp/cancer free, pre-cancerous and confirmed primary diagnosis of colorectal cancer (stage I, II and III) will be recruited. Participants will be recruited in primary, secondary, and tertiary care centers, depending on the study inclusion/exclusion criteria.

Participants complete surveys and collect samples including (blood, urine, stool, and saliva) using at-home/in-clinic kits provided by Viome. Participants are also asked to provide tissue or tumor samples if collected by their healthcare provider during a standard of care biopsy procedure. Biopsy samples for this test will be collected by the clinical staff at each study site. Additional data collection, including medical data, biopsies and other biological samples might happen at interim timepoints in case of adenoma/cancer disease progression (recurrence, metastasis). Additionally, participants complete a survey sent on a quarterly basis.

There are 5 timepoints (TP) in this study including: Timepoint 1, Timepoint 2, Timepoint 3, Timepoint 4, and Timepoint 5.

TP1 includes the initial diagnosis where the stage of cancer is determined by imaging (colorectal cancer stages I, II, or III) or colonoscopy results (healthy and pre-cancerous). All participants provide urine, blood, saliva, stool and complete survey.

TP2 includes Post Standard of Care (SOC). For cancer participants, samples will be collected 45 +/- 15 days after all treatments have been completed (this includes chemotherapy, radiation therapy, immunotherapy, and/or surgery). Those that are healthy and pre-cancerous will provide their samples, 90 +/- 15 days after the colonoscopy. All participants provide urine, blood, saliva, stool and complete survey.

TP3, 4, and 5 occur 1, 2 and 3 years respectively after diagnosis (TP1) for cancer-free and precancerous groups and 1, 2 and 3 years respectively after standard of care therapy (TP2) for the cancer groups. All participants provide urine, blood, saliva, stool and complete survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* with a signed Informed Consent Form
* able to comply with the protocol requirements AND
* Confirmed primary diagnosis of colorectal cancer (stage I (1), II (2) and III (3)), or pre-- cancerous polyps, including tubulovillous or villous adenomas, with a biopsy available for study assays OR
* CRC-free and polyp-free colon using colonoscopy

Exclusion Criteria:

* Diagnosis of CRC relapse at the time of enrollment
* Inflammatory bowel disease
* Irritable bowel syndrome (IBS), confirmed at enrollment
* Pregnant, planning to become pregnant during the study timeline or nursing
* Cholecystectomy (gallbladder removal)
* Bariatric/gastric surgery
* Partial colectomy (colon removal)
* Partial bowel resection
* Pancreatic surgery
* Lynch syndrome
* Familial polyposis
* Patients from which the healthcare providers do not collect biopsy at colonoscopy AND undergo neoadjuvant therapy prior to surgery (the microbial composition of the biopsy at the time of surgery may be significantly affected by neoadjuvant therapy).
* Known autoimmune condition or impairment of immunological functions (e.g. HIV infection)
* Medications: Receipt of biologics, systemic immunosuppressive therapy, incl. cancer therapy, or antibiotics in the last 3 months before initial diagnosis
* Any vaccine taken within the last 30 days
* Current receipt of investigational agent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited into the following study groups:
  Cancer-free subjects (confirmed CRC-free via colonoscopy) Precancerous stage participants Stage I (1) colorectal cancer participants Stage II (2) colorectal cancer participants Stage III (3) colorectal cancer participants
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
The molecular features of Fusobacterium (Fn) correlated with colorectal cancer (onset, recurrence, metastasis and survival) | 6 years
  Determine Fn species and strains, more specifically the prevalence and relative activity, and the differential gene expression and key pathways. The Investigators will also look at Microbial co-occurrence/abundance with Fn and local tumor microenvironment and tumor marker/mutations and their association with microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, PhD, Principal Investigator — Viome
Locations (1):
- Washington Gastroenterology, Bellevue, Washington, United States